CLINICAL TRIAL: NCT04934618
Title: A Single-arm, Multicenter, Open-labeled, Phase II Study on the Efficacy and Safety of Carelizumab Combined With Irinotecan and Apatinib in the Second-line Treatment of Locally Advanced Unresectable, Recurrent or Metastatic Adenocarcinoma of Stomach and Gastroesophageal Junction
Brief Title: A Phase II Study of Carelizumab Combined With Irinotecan and Apatinib of Second-line Treatment for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Shimin, Vice director of Oncology Department, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2020-024
Record Dates: First submitted 2021-06-12; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carelizumab Combined With Irinotecan and Apatinib (Experimental): Second-line treatment of advanced gastric cancer with three-drug regimen（Carelizumab Combined With Irinotecan and Apatinib ）
  Interventions: Drug: Carelizumab Combined With Irinotecan and Apatinib

INTERVENTIONS:
Drug: Carelizumab Combined With Irinotecan and Apatinib — Three-drug regimen was used in second-line treatment of Advanced gastric cancer

SUMMARY:
The purpose of this study was to evaluate the overall survival time (OS), objective remission rate（ORR）, progression-free survival time（PFS）, disease control rate（DCR）of Carelizumab combined with irinotecan and apatinib for the second-line treatment of locally advanced unresectable, recurrent or metastatic adenocarcinoma of stomach and gastroesophageal junction. At the same time, the safety and tolerance of the scheme were preliminarily evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. The local advanced stage confirmed by histopathology is unresectable, recurrent or metastatic Adenocarcinoma of stomach and gastroesophageal junction.
2. After receiving first-line treatment, the disease progressed or intolerable adverse reactions occurred.
3. At least one measurable lesion or evaluable lesion (according to RECIST 1.1 standard);
4. Patients agreed to provide blood samples and previously stored tumor tissue samples for tumor microenvironment detection.
5. Age ≥18 years old and ≤75 years old.
6. The ECOG score is 0 or 1.
7. The estimated survival time is ≥3 months.
8. Within 7 days before entering the group, the laboratory test value met the chemotherapy standard.
9. Within 28 days before enrollment, women of childbearing age must confirm that the serum pregnancy test is negative and agree to adopt effective contraceptive measures during the study drug use and within 6 months after the last administration.
10. Patients voluntarily joined the study, signed informed consent, and were able to comply with the visit and related procedures stipulated in the plan.

Exclusion Criteria:

1. Participate in other intervention clinical studies at the same time (unless participating in observation studies or being in the follow-up stage of intervention studies), and have received second-line treatment.
2. have received antibody therapy of PD-1, PD-L1, PD-L2, CTLA4, CD137 or any other antibody or drug therapy with t cell co-stimulation or immune checkpoint pathway as specific target.
3. It is known to be allergic to any monoclonal antibody or adjuvant.
4. Received Chinese patent medicines with anti-tumor indications or drugs with immunoregulatory effects (thymosin, interferon, interleukin, etc.) within 2 weeks before the first administration.
5. Having undergone major surgery within 4 weeks before the first administration or expecting to undergo surgery during the study treatment.
6. Receive live attenuated vaccine within 4 weeks before the first administration or during the planned study treatment.
7. Received transplantation of solid organs or blood system.
8. Active, known or suspected autoimmune diseases or related medical history in the past 2 years (vitiligo, psoriasis, alopecia or Graves' disease that does not require systematic treatment in the past 2 years, hypothyroidism that only requires thyroid hormone replacement therapy, and type I diabetes patients who only need insulin replacement therapy can enter Group).
9. Immunosuppressive drugs have been used within 4 weeks before the first administration, excluding local glucocorticoid by nasal spray, inhalation or other routes or systemic glucocorticoid with physiological dose (i.e., prednisone or other glucocorticoid with equivalent dose not exceeding 10mg/ day), or hormone used due to allergy.
10. Known history of primary immunodeficiency disease.
11. Known history of active tuberculosis. 12 known to have a history of human immunodeficiency virus (HIV) infection (i.e., HIV antibody positive).

13. after regular antihypertensive treatment, the blood pressure still cannot fall to the normal range (systolic blood pressure > >140mmHg, diastolic blood pressure > >90mmHg).

14. ≥II grade ii coronary heart disease and arrhythmia (including QTc interval prolongation > >450ms for men and > >470ms for women).

15. Symptomatic congestive heart failure (new york Heart Association Grade II-IV) or symptomatic or poorly controlled arrhythmia.

16. before the first administration, there was toxicity caused by previous anti-tumor treatment that did not recover to grade 0 or grade 1 of the national cancer institute general adverse event terminology version 4.03 (NCI ctcae version 4.03) (excluding alopecia, fatigue and asymptomatic laboratory abnormalities).

17. abnormal coagulation function (INR > 1.5 uln, aptt > 1.5 uln), with bleeding tendency.

18. It is known that symptomatic central nervous system metastasis exists. 19. Diagnosed as other malignant tumors within 5 years before the first administration, excluding basal cell carcinoma of skin, squamous cell carcinoma of skin and carcinoma in situ after radical resection.

20. Active infections requiring treatment or systemic anti-infective drugs used within 7 days before the first administration.

21. acute or chronic active hepatitis b: HBV viral load ≥500 copies /ml 22. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before the study.

23. It is known that there are mental diseases or drug abuse situations that may affect the compliance with the test requirements.

24. Acute or chronic active hepatitis C: HCV antibody is positive. 25. Pregnant or lactating women. 26. There are medical histories, diseases, treatments or abnormal laboratory results that may interfere with the test results and prevent the subjects from participating in the study, or the researchers think that participating in the study is not in the best interests of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2020-05-19 (Actual); Primary Completion 2023-05-19 (Estimated); Study Completion 2025-05-19 (Estimated)

PRIMARY OUTCOMES:
Overall Suvival time（OS） | Up to 24 months
  The time from randomization to death due to any reason. For those who have lost follow-up before death, the last follow-up time is usually calculated as the time of death.

SECONDARY OUTCOMES:
Progress Free Survival time（PFS） | Up to 24 months
  The time from randomization to the first occurrence of disease progression or death from any cause.
objective response rate（ORR） | Up to 24 months
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and kept for a certain time, including CR and PR cases
duration of response （DoR） | Up to 24 months
  It is the curative effect evaluation index of tumor reaction, which refers to the time from the first evaluation of complete remission (CR) or partial remission (PR) to the first evaluation of disease progression (PD) or death from any cause
Disease control rate（DCR） | Up to 24 months
  The proportion of patients whose tumors have shrunk or remained stable for a certain period of time, including cases of complete remission (CR), partial remission (PR) and stable (SD)

OTHER OUTCOMES:
Safety and tolerability | Up to 24 months
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Min Shi, Principal Investigator — Oncology department of Nanfang hospital
Locations (1):
- NanFang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No